CLINICAL TRIAL: NCT00979823
Title: Simulated Diabetes Training for Resident Physicians
Acronym: SDT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HealthPartners Institute (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: X0710100 Resident SimCare; R18DK079861 (NIH)
Record Dates: First submitted 2009-09-16; First posted 2009-09-18 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-12

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early SimCare Diabetes Group (Experimental): This group will receive an email web-link to 3 simulated learning cases each month for 6 months. After 6 months (18 total learning cases), they will then complete 4 simulated assessment cases, a diabetes knowledge survey, and a satisfaction survey.
  Interventions: Other: Early SimCare Diabetes Group
- Delayed SimCare Diabetes Group (Active Comparator): Beginning in the spring of 2011, residents in this group will receive an email web-link to complete 4 simulated assessment cases and a diabetes knowledge survey. They will subsequently be sent 3 learning cases a month for 6 months and a satisfaction survey to complete.
  Interventions: Other: Delayed SimCare Diabetes Group

INTERVENTIONS:
Other: Early SimCare Diabetes Group — Residents in the early learning program group will participate in the learning cases before undergoing a knowledge and performance assessment. They will complete 18 learning cases, 4 assessment cases, knowledge survey, and a satisfaction survey.
  Arms: Early SimCare Diabetes Group
Other: Delayed SimCare Diabetes Group — Residents in the delayed learning program group will receive their usual diabetes training through their residency program for 8 months before completing the knowledge and performance assessment, and then will subsequently be offered the learning program. They will receive 4 assessment cases, knowledge survey, and satisfaction survey
  Arms: Delayed SimCare Diabetes Group

SUMMARY:
The objective of this translational research is to study the effect of implementing an innovative simulated diabetes learning intervention within primary care residency programs. The intervention uses cognitive behavioral learning theory to provide goal-directed feedback to residents after every encounter over a series of virtual patient-physician encounters. Formulas derived from pharmacokinetic data and the experience of clinical experts model simulated physiologic responses to drug changes, health behaviors, and adherence factors. The online intervention is economical, sustainable, and addresses a number of current obstacles to outpatient diabetes training in primary care residency programs.

In this group trial, we randomly assign about 20 primary care residency programs with up to 700 residents total to either an (a) Early learning program group or (b) Delayed learning program group. We will assess the ability of residents to achieve evidence-based diabetes clinical goals and avoid potential medical safety issues for glycemia, blood pressure, and lipids on simulated assessment cases. Secondary analyses will evaluate the actual use of the tool by residents, direct costs of the program, and resident satisfaction.

DETAILED DESCRIPTION:
Specific aim 1: To examine the impact of a simulated case-based learning intervention on measures of quality of diabetes care delivered by primary care residents to simulated adult patients with diabetes mellitus.

Hypothesis 1: Compared to delayed SimCare Diabetes learning program group residents, those residents in the early SimCare Diabetes learning program group will treat a higher proportion of simulated patients to evidence based diabetes goals including glycemic control (A1c < 7%), blood pressure control (BP < 130/80 mm Hg), and lipid control (evidence-based LDL, Triglyceride, and HDL levels).

Specific aim 2: To examine the impact of a simulated case-based learning intervention on rates of appropriate drug intensification and number of risky prescribing events in the management of simulated adult patients with diabetes mellitus.

Hypothesis 2: Compared to delayed SimCare Diabetes learning program group residents, those residents in the early SimCare Diabetes learning program group will have improved rates of appropriate drug intensification in simulated assessment cases.

Hypothesis 3: Compared to delayed SimCare Diabetes learning program group residents, those residents in the early SimCare Diabetes learning program group will have a lower number of risky prescribing events in simulated assessment cases.

ELIGIBILITY:
Study subjects include up to 700 first, second, third, and fourth year primary care residents from a minimum of 20 residency programs across the country. To become a partner in this study, programs must meet the eligibility criteria listed below:

To be eligible for partnership in this study, a program must meet all the following criteria:

a) be an accredited family medicine or internal medicine/med-peds training program within the U.S., (b) have a minimum of 12 residents within the standard 3- to 4-year program, (c) the program director must endorse and be willing to offer SimCare Diabetes to all residents within the program and provide residents (with help from the study staff) with the explanatory and registration materials, (d) the residency program director must sign a letter of agreement with the research team specifying the responsibilities of the research team and of the residency program in addressing the specific needs of this project, (e) the residency program director must agree to complete a residency program director survey, which provides insight into the general characteristics of the residency program, and provide diabetes quality measurement data from at least one resident ambulatory clinic pre-intervention (around October/November 2010) and post-intervention (around June/July 2011), (f) residents within the program must have high speed internet access, and (g) if randomized to the delayed learning program group, the program must be willing to postpone SimCare Diabetes until after the post-intervention assessment cases are completed.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2010-09; Primary Completion 2012-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Treatment according to evidence-based diabetes goals | September 2010 - July 2013
Drug intensification | September 2010 - July 2013
Number of risky prescribing events | September 2010 - July 2013

SECONDARY OUTCOMES:
Secondary analyses will evaluate the actual use of the tool by residents, direct costs of the program, and resident satisfaction. | July 2011 - January 2013

CONTACTS AND LOCATIONS:
Overall Officials: JoAnn M Sperl-Hillen, MD, Principal Investigator — HealthPartners Institute
Locations (1):
- HealthPartners Research Foundation, Minneapolis, Minnesota, United States

REFERENCES:
- [Derived] Sperl-Hillen JM, O'Connor PJ, Rush WA, Johnson PE, Gilmer T, Biltz G, Asche SE, Ekstrom HL. Simulated physician learning program improves glucose control in adults with diabetes. Diabetes Care. 2010 Aug;33(8):1727-33. doi: 10.2337/dc10-0439. PMID 20668151